CLINICAL TRIAL: NCT03376776
Title: Epiretinal Proliferation in Eyes With Full Thickness Macular Hole
Status: Completed | Type: Observational
Sponsor: Kyorin University (Other)
Responsible Party: Principal Investigator, Makoto Inoue, Professor of Ophthalmology, Kyorin University
Other Study IDs: Kyorineye024
Record Dates: First submitted 2017-12-13; First posted 2017-12-18 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Macular Disease
Keywords: idiopathic macular hole
MeSH Terms: conditions — Macular Degeneration | interventions — Vitrectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Eyes with epiretinal proliferation: The eyes with epiretinal proliferation around the macular hole detected with optical coherence tomography
  Interventions: Procedure: Vitrectomy
- Eyes without epiretinal proliferation: The eyes without epiretinal proliferation around the macular hole detected with optical coherence tomography
  Interventions: Procedure: Vitrectomy

INTERVENTIONS:
Procedure: Vitrectomy

SUMMARY:
We evaluated preoperative and postoperative optical coherence tomograpghic images in eyes with full thickness macular hole (FTMH) whether the epiretinal proliferation (EP) was detected and detection of EP was correlated to the visual improvement.

DETAILED DESCRIPTION:
We evaluated preoperative and postoperative optical coherence tomograpghic images in eyes with full thickness macular hole (FTMH) whether the epiretinal proliferation (EP) was detected and detection of EP was correlated to the visual improvement.

ELIGIBILITY:
Inclusion Criteria:

* Eyes with macular hole

Exclusion Criteria:

* Eyes with retinal detachment, retinal vascular disease, glaucoma, proliferative diabetic retinopathy

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The eyes with macular hole
Sampling Method: Probability Sample
Enrollment: 390 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Recovery of foveal microstructure | 6 months

SECONDARY OUTCOMES:
Visual improvement | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Makoto Inoue, MD, Principal Investigator — Kyorin Eye Center
Locations (1):
- Makoto Inoue, Mitaka-shi, Tokyo, Japan